CLINICAL TRIAL: NCT05576155
Title: Sex Differences in the Dilatory Response of Compound 21
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202206519
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Sex Differences
MeSH Terms: interventions — compound 21; Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Local losartan perfusion (Experimental): ~1 hour of losartan is perfused through an intradermal microdialysis fiber
  Interventions: Drug: Compound 21 + losartan
- Local lactated Ringer's (control) perfusion (Other): ~1 hour of lactated Ringer's is perfused through an intradermal microdialysis fiber
  Interventions: Drug: Compound 21

INTERVENTIONS:
Drug: Compound 21 — Compound 21 + Ringer's is perfused at 10 doses increasing serially for 10 minutes each from 10^-12 M to 10^-3 M
  Arms: Local lactated Ringer's (control) perfusion
Drug: Compound 21 + losartan — Compound 21 + losartan (43 µM) is perfused at 10 doses increasing serially for 10 minutes each from 10^-12 M to 10^-3 M.
  Arms: Local losartan perfusion

SUMMARY:
When blood pressure changes, Angiotensin II is produced and released into the bloodstream. This substance can make blood vessels smaller (i.e., vasoconstriction) by acting through Angiotensin II type I receptors (AT1R) to increase blood pressure. Or it can increase the diameter of vessels (i.e., vasodilation) through Angiotensin II type II receptors (AT2R) to decrease blood pressure. These two receptors normally work in balance to maintain blood pressure. However, excess Angiotensin II released in the bloodstream may reduce the sensitivity of AT2Rs, leading to excessive activation of AT1Rs. This results in increased constriction which plays a major role in diseases such as high blood pressure, hardening of the arteries, and heart failure. In the body, Angiotensin II production is reduced in the presence of estrogen, as seen in pre-menopausal women. Pre-menopausal women have a greater protection against cardiovascular diseases compared to age-matched males, likely due to the protective effects of estrogen. However, the extent that estrogen may impact the sensitivity of Angiotensin II receptors in pre-menopausal is unknown.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents), the blood vessels in a dime-sized area of the skin are studied in healthy young women and men. As a compliment to these measurements, blood is drawn from the subjects and circulating factors that may contribute to cardiovascular health are measured.

ELIGIBILITY:
Inclusion Criteria:

* Young women or men,
* 18-35 years old,
* Body mass index between 18 and 30 kg/m2,
* Systolic blood pressure <140,
* Diastolic blood pressure <90 mmHg.

Exclusion Criteria:

* Skin allergies, skin disorders, or skin diseases such as Raynaud's phenomenon or other history of cold intolerance,
* History of metabolic or cardiovascular disease,
* Taking medications that could alter vascular function, including antidepressants, anxiety medications, or cholesterol or blood pressure lowering drugs,
* Women with oligo- or amenorrhea,
* Women that are pregnant or nursing
* current tobacco use,
* Allergy to materials used during the experiment (e.g. latex).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Men: Young men aged 18-35
- Young Women: Premenopausal women aged 18-35
Period: Overall Study
Arm/Group | Young Men | Young Women
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Men | Young Women | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (5) | 22 (3) | 22 (24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 12
  Male | 12 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Heart rate [Mean (Standard Deviation); unit: bpm] | 59 (11) | 64 (11) | 62 (11)
Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 82 (6) | 79 (6) | 80 (6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25 (2) | 24 (2) | 24 (2)

OUTCOME MEASURES:

1. Primary Outcome: Microvascular AT2R Sensitivity Following Local Control Treatment
Description: cutaneous vascular vasodilator response to exogenous Compound 21 perfusion; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of Compound 21 in young men and women
Time Frame: post 1 hour of local control treatment
Measure: Mean (Standard Error); unit: percentage of maximal blood flow
Arm/Group | Young Men | Young Women
Number analyzed (Participants) | 12 | 12
percentage of maximal blood flow | 15 (2) | 25 (4)

2. Primary Outcome: Microvascular AT2R Sensitivity Following Local AT1R Inhibition
Description: cutaneous vascular vasodilator response to exogenous Compound 21 perfusion; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of Compound 21 co-infused with losartan young men and women
Time Frame: post 1 hour of local losartan treatment
Measure: Mean (Standard Error); unit: percentage of maximal blood flow
Arm/Group | Young Men | Young Women
Number analyzed (Participants) | 12 | 12
percentage of maximal blood flow | 26 (4) | 27 (6)

3. Secondary Outcome: Circulating Progesterone and Testosterone
Description: plasma measurement of circulating progesterone and testosterone; measured by ELISA in plasma samples
Time Frame: at the start of the experimental visit, immediately prior to local losartan treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Young Men | Young Women
Number analyzed (Participants) | 10 | 8
ng/mL
  Progesterone | 0.9 (0.8) | 0.7 (0.4)
  Testosterone | 1029.4 (556.1) | 174.1 (97.4)

4. Secondary Outcome: Circulating Estradiol
Description: plasma measurement of circulating estradiol, measured by ELISA in plasma samples
Time Frame: at the start of the experimental visit, immediately prior to local losartan treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Young Men | Young Women
Number analyzed (Participants) | 10 | 8
pg/mL | 134.1 (83.4) | 138.5 (133.1)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Monitored through study completion
Arm/Group | Young Men | Young Women
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT05576155/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT05576155/ICF_001.pdf